CLINICAL TRIAL: NCT01389479
Title: Active-control Study to Evaluate the Safety, Tolerance and Immunogenicity of Fluviral™ S/F Influenza Vaccine in Healthy Adults Aged 18-64 Years of Age
Brief Title: Study to Evaluate the Safety, Tolerance and Immunogenicity of Fluviral™ in Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: ID Biomedical Corporation, Quebec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IDB-707-105
Record Dates: First submitted 2011-07-04; First posted 2011-07-08 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

ARMS (2):
- Fluviral Group (Experimental)
  Interventions: Biological: Fluviral™
- Fluzone Group (Active Comparator)
  Interventions: Biological: Fluzone®

INTERVENTIONS:
Biological: Fluviral™ — Intramuscular, single dose
  Arms: Fluviral Group
Biological: Fluzone® — Intramuscular, single dose
  Arms: Fluzone Group

SUMMARY:
The purpose of the study is to evaluate the safety, tolerance and immunogenicity of Fluviral™ in healthy adults aged 18-64 years.

DETAILED DESCRIPTION:
This study was conducted by ID BioMedical which has been taken over by GlaxoSmithKline. At the time of conduct of this study, Fluviral was produced by ID BioMedical.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Adults 18-64 years of age, inclusive.
* Satisfactory baseline medical assessment by history, physical examination, and clinical laboratory testing.
* Capable of informed consent.
* Able, willing and likely to fully comply with study procedures and restrictions.

Exclusion Criteria:

* Acute illness at the time of enrollment.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus infection and/or chronic use of immunosuppressants of other immune-modifying drugs within 6 months of administration of the study vaccine.
* Presence of an unstable chronic illness.
* Complicated diabetes mellitus.
* Active neurological disorder.
* History of any demyelinating disease including Guillain-Barré syndrome.
* Any clinical laboratory abnormality.
* Any disorder of coagulation or treatment with coumadin derivatives or heparin.
* Vital sign abnormalities at screening.
* Acute or chronic liver, renal or inflammatory bowel disease or collagen vascular disease.
* Cancer, or treatment for cancer, within three years.
* History of significant alcohol or drug abuse within one year prior to the screening visit.
* Positive urine drug screen at screening within 3 months prior to the screening visit or hard drugs. Products such as ativan, tylenol with codeine should be stopped sufficiently ahead of the screening visit in order to avoid a positive urine drug screen.
* Positive testing for hepatitis B, hepatitis C or human immunodeficiency virus at screening.
* Receipt of an influenza vaccine within 9 months prior to dosing.
* Planned administration of any other vaccines 30 days before study immunization or during the course of the study. Immunization on an emergency basis, such as Tetanus and Diphtheria Toxoids Adsorbed for adult use, will be allowed provided the vaccine is not administered within two weeks prior to study immunization.
* Use of any investigational or non-registered drug or vaccine or participation in an investigational study within 30 days prior to administration of study vaccine, or planned use during the study period.
* Receipt of any immunoglobulins and/or any blood products within three months of screening or planned administration of any of these products during the study period.
* Receipt of a depot injection or an implant of any drug within 3 months prior to administration of study vaccine.
* Any known or suspected allergy to any constituent of Fluviral™ S/F or Fluzone®.
* A history of severe adverse reaction to a previous dose of any influenza vaccine.
* History of anaphylactic type reactions to consumption of eggs.
* Any other condition or social circumstance that, in the opinion of the Principal Investigator, would make the subject unsuitable for or unable to complete the study.
* Breast-feeding subject.
* Positive urine pregnancy test at screening.
* Female subjects having sexual intercourse with any non-sterile male partner within 14 days prior to vaccine administration and without a history of acceptable contraception.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1000 (Actual)
Dates: Start 2005-01; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects with solicited local and systemic reactogenicity symptoms | First three days after vaccination
Number of subjects reporting spontaneous adverse events | Throughout the entire study period (Day 0-42)
Immune response in terms of number of seroconverted subjects | Before (Day 0) and after (Day 21) vaccination
Immune response in terms of number of seroprotected subjects | Before (Day 0) and after (Day 21) vaccination

SECONDARY OUTCOMES:
Immunogenicity with respect to components of the study vaccine in terms of number of subjects with titres above the pre-defined cut-off | At Day 21 after vaccination
  Titres calculated as geometric mean
Immune response to components of the study vaccine in terms of mean Geometric increase | At Day 21 after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline